CLINICAL TRIAL: NCT03163641
Title: A Randomized, Masked (Reading Center), Prospective Pilot Study of the Safety and Effectiveness of the EyeGate Ocular Bandage Gel, a 0.75% Crosslinked Hyaluronic Acid Applied Topically, Versus a Bandage Contact Lens for Acceleration of Re-epithelialization of Large Corneal Epithelial Defects in Patients Having Undergone Photorefractive Keratectomy (PRK).
Brief Title: Safety and Effectiveness of OBG vs.a Bandage Contact Lens for Large Corneal Epithelial Defects in Patients Post-PRK.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eyegate Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EYEGATE-033
Record Dates: First submitted 2017-05-17; First posted 2017-05-23 (Actual); Last update posted 2020-12-17 (Actual); Status verified 2019-01

CONDITIONS: Corneal Epithelial Wound
Keywords: Photorefractive Keratectomy, Corneal Defect

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Used a masked reading center to review the corneal defect staining.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (3):
- Treatment 1 (Experimental): Ocular Bandage Gel
  Interventions: Device: Ocular Bandage Gel
- Treatment 2 (Experimental): Ocular Bandage Gel
  Interventions: Device: Ocular Bandage Gel
- Control Group (Active Comparator): Artificial tears with Acuvue Oasys
  Interventions: Device: Acuvue Oasys; Device: Ocular Bandage Gel

INTERVENTIONS:
Device: Acuvue Oasys — Bandage Contact Lens
  Arms: Control Group
Device: Ocular Bandage Gel — 0.75% crosslinked HA

SUMMARY:
This is a prospective, randomized (Reading Center), masked, controlled study in up to 45 subjects who have undergone bilateral PRK with epithelial removal using alcohol in a 9.0 mm well or trephine at the time of surgery to ensure consistency of the size of the ablation area.

DETAILED DESCRIPTION:
This is a prospective, randomized (Reading Center), masked, controlled study in up to 45 subjects who have undergone bilateral PRK with epithelial removal using alcohol in a 9.0 mm well or trephine at the time of surgery to ensure consistency of the size of the ablation area. Subjects will be assigned to one of three treatment arms on Day 0.

ELIGIBILITY:
Inclusion Criteria:

* Able and willing to comply with the protocol

Exclusion Criteria:

-

Ages: 22 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2018-08-05 (Actual); Primary Completion 2018-10-31 (Actual); Study Completion 2018-11-08 (Actual)

PRIMARY OUTCOMES:
Time to corneal re-epithelization post PRK | Day 3
  Time to corneal re-epithelization post PRK

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Wirostko, M.D., Study Director — Eyegate Pharmaceuticals, Inc.
Locations (1):
- Houston, Texas, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Durrie DS, Wolsey D, Thompson V, Assang C, Mann B, Wirostko B. Ability of a new crosslinked polymer ocular bandage gel to accelerate reepithelialization after photorefractive keratectomy. J Cataract Refract Surg. 2018 Mar;44(3):369-375. doi: 10.1016/j.jcrs.2018.01.018. PMID 29703289